CLINICAL TRIAL: NCT02249702
Title: A Phase II Randomized - Non Comparative - Study on the Activity of Trabectedin or Gemcitabine + Docetaxel in Metastatic or Locally Relapsed Uterine Leiomyosarcoma Pretreated With Conventional Chemotherapy
Brief Title: Activity of Trabectedin or Gemcitabine + Docetaxel in Uterine Leiomyosarcoma
Acronym: TAUL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAUL; 2009-016017-24 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Leiomyosarcoma
Keywords: trabectedin; uterine leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Gemcitabine; Docetaxel; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabectedin (Experimental): Trabectedin 1.3 mg/m2 will be administered via a central venous catheter as a 24-hour infusion on day 1 of 21-days treatment cycles. Trabectedin treatment can be continued until progressive disease, major toxicity, patient's intolerance or unwillingness to continue treatment or medical decision by the responsible physician.
  Interventions: Drug: trabectedin
- gemcitabine + docetaxel (Active Comparator): Gemcitabine 900 mg/m2 will be administered via a central venous catheter on days one and eight over 90 min, followed by docetaxel 75 mg/m2 on day eight iv over 1 h. Gemcitabine+docetaxel treatment is planned for six cycles, unless there is evidence of disease progression, unacceptable toxicity or patient's intolerance or unwillingness to continue treatment, or medical decision by the responsible physician. Patients with continued response after six cycles can receive two additional cycles of combination therapy or continue with Gemcitabine alone.
  Interventions: Drug: gemcitabine + docetaxel

INTERVENTIONS:
Drug: gemcitabine + docetaxel
  Other Names: Gemzar; Taxotere
  Arms: gemcitabine + docetaxel
Drug: trabectedin
  Other Names: Yondelis
  Arms: Trabectedin

SUMMARY:
The management of patients with uterine leiomyosarcomas poses many difficulties. Despite 60% of women present with disease limited to the uterus, cure rates range from 20 to 60%. Patients with metastatic disease at diagnosis or who recur after initial treatment have a dismal prognosis and, except for a subset of selected patients with completely resectable disease, the median survival is less than one year. Treatment options for recurrent/metastatic uterine leiomyosarcoma are limited. The most active drugs are doxorubicin ± ifosfamide and gemcitabine + docetaxel (GD) with response rate of 25-55% and 27-53%, respectively. Both these regimens have been increasingly used in the last years also in the adjuvant setting. For relapsed patients other drugs have been tested as single agent but negligible activity was observed.

Trabectedin (Yondelis® -T) is a marine-derived cytotoxic approved by EMEA. It is indicated for the treatment of patients with advanced soft tissue sarcoma, after failure of anthracyclines and ifosfamide or who are unsuitable to receive these agents. Among STS, activity has been mainly detected in synovial sarcoma, liposarcoma and leiomyosarcoma. Although the response rate did not exceed 10%, T was demonstrated to provide disease control, with progression arrest rates exceeding 50% and progression-free survival rates exceeding 20% at 6 months. So far no phase II studies tested the activity of T in uterine leiomyosarcoma specifically. This study is aimed at evaluating the activity of T (arm A) in advanced uterine leiomyosarcomas, having GD (arm B) as an internal control In parallel translational studies will be performed to identify factors predictive of the activity of T in this specific histotype.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven uterine leiomyosarcoma.
2. Persistent or locally relapsed and/or metastatic disease.
3. At least one previous systemic treatment with an anthracycline ± ifosfamide or gemcitabine ± docetaxel.
4. Measurable disease, as defined by RECIST criteria.
5. ECOG PS <=2.
6. Age >= 18 years.
7. A minimum of 3 weeks since prior tumor directed therapy
8. Recovery from toxic effects of prior therapies to NCI CTC Grade 1 or lower.
9. Adequate haematological function.
10. Adequate renal function.
11. Adequate liver function.
12. Signed informed consent.

Exclusion Criteria:

1. Prior exposure to Trabectedin.
2. Peripheral neuropathy, Grade 2 or higher.
3. History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission from 5 years or more and judged of negligible potential of relapse.
4. Known CNS metastases.
5. Active viral hepatitis or chronic liver disease.
6. Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within one year before enrolment, uncontrolled arterial hypertension or arrhythmias.
7. Active major infection.
8. Other serious concomitant illnesses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-04; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
progression free rate at 6-month | 6-month
  Primary objective will be to assess the clinical benefit rate (defined as 6-month progression free rate) with trabectedin in patients with locally relapsed/metastatic uterine leiomyosarcoma pretreated with anthracycline ± ifosfamide and/or gemcitabine ± docetaxel.

SECONDARY OUTCOMES:
best response rate | within 6 months
  response rate according to RECIST v1.0 criteria

OTHER OUTCOMES:
progression free survival | 24 months
  Time from inclusion into the study to progression or death whichever comes first
Overall survival | 24 months
  time from inclusion into the study to death from any cause
safety profile | up to 30 days after the end of treatments
  Number of Patients with Serious and Non-Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Angiolo Gadducci, MD, Principal Investigator — Azienda Ospedaliero Universitaria Pisana, Pisa, Italy; Federica Grosso, MD, Principal Investigator — Azienda Ospedaliera Alessandria, Italy
Locations (33):
- Italy (33):
  - Centro di Riferimento Oncologico, Aviano, Pordenone
  - Policlinico Umberto I, Roma, RM
  - Fondazione del Piemonte per l'Oncologia, Candiolo, Turin
  - Azienda ULSS 13 Regione Veneto, Ospedale di Mirano, Mirano, Venice
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Presidio Ospedaliero Senatore Antonio Perrino, Brindisi
  - Azienda Ospedaliera per l'Emergenza Cannizzaro, Catania
  - Ospedale Sant'Anna, Como
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Azienda Ospedaliera Universitaria San Martino - IST, Genoa
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Azienda USL 2 Toscana - Nuovo Ospedale San Luca, Lucca
  - Istituto Clinico Humanitas, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale dei Tumori di Milano, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Istituto Nazionale Tumori - Fondazione Pascale, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Policlinico San Matteo, Pavia
  - Azienda Ospadaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliera Regionale San Carlo, Potenza
  - Azienda Ospedaliera Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Umberto I - Università Sapienza, Roma
  - Policlinco Universitario Agostino Gemelli, Rome
  - Azienda Ospedaliera Ordine Mauriziano, Torino
  - Azienda Ospedaliero-Universitaria di Torino - Presidio Sant'Anna, Torino
  - Presidio Sanitario Gradenigo, Torino